CLINICAL TRIAL: NCT03397017
Title: National Transfusion Treatment Survey in Patients With Sickle Cell Disease (SCD)
Brief Title: Transfusion Treatment in Patients With SCD
Status: Completed | Type: Observational
Sponsor: Società Italiana Talassemie ed Emoglobinopatie (Other)
Collaborators: Associazione Italiana de Ematologia e Oncologia Pediatrica (Unknown); Società Italiana di Medicina Trasfusionale e Immunoematologia (Unknown)
Responsible Party: Sponsor
Other Study IDs: SITE
Record Dates: First submitted 2017-12-18; First posted 2018-01-11 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Anemia, Sickle Cell
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Blood Transfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Transfusion

SUMMARY:
The "National Transfusion Treatment Survey in patients with sickle cell disease (SCD)" is a prospective longitudinal systemic study that was created in order to evaluate the therapeutic approach, mainly transfusional, in patients affected by SCD throughout Italy and to improve the quality of care and implement research.

The survey will evaluate all patients affected by different forms of sickle cell disease (HbS homozygosis, Thalassoso-drepanocytosis, HbS / HbC compound heterozygosis, other possible genetic compounds).

Patients will be selected according with a SCD diagnosis confirmed by standardized biochemical criteria or by DNA analysis. Patients will be excluded from the study who do not meet the these requirements, who are unable to understand the protocol or able to give informed consent in the absence of any legal representative.

All data will be collected through a standard web-based application, which will be completed by the responsable investigator or by sub-investigators selected by each center, after registration on the site providing personal data and indicating the affiliation structure. All data will be subsequently encrypted by the Central Server. The operator will subsequently be able to access the patient's clinical data to perform the updates, in order to follow the patient's clinical evolution over time. The study will not involve any additional tests compared to the routine of patient control.

DETAILED DESCRIPTION:
Sickle Cell Disease (SCD) includes a group of rare inherited monogenic diseases caused by mutations of genes involved in hemoglobin biosynthesis and is characterized by the presence of a hemoglobin variant (HbS); transmission occurs according to mendelian recessive mode.

The term "Sickle Cell Disease" includes several genotypes expressing a similar phenotype, characterized by acute events sustained from the pathophysiological point of view by vasoocclusive and / or acute hemolytic crisis and by chronic hemolytic anemia, mechanisms both conditioning in progressive organ damage time. The most common genotype (70% present in the African continent) consists of homozygosity for both alleles S (Drepanocytosis or Sickle Cell Anemia, SCA - HbSS), followed by compound heterozygosis of a β-thalassemic mutation and an allele S ( Thalasso-sickle cell disease or HbS / βthal), then from βs/ βc (HbS / HbC hemoglobinopathy).

The characteristic clinical manifestations consist of recurrent vaso-occlusive ischemic events and consequent micro infarcts, up to the development of acute and chronic multi-organ insufficiency; the responsible pathophysiological mechanism resides in the polymerization of hemoglobin S.

The main acute, life-threatening events are acute cerebrovascular events (stroke, 11% of patients with SCA within 20 years), acute respiratory failure (Acute Chest Syndrome, ACS) associated with pulmonary hypertension and severe painful osteo-articular and splanchnic crises.

The identification and detection of parameters indicating the progressive deterioration of neurological and cardio-pulmonary function could be decisive in the prevention of both acute events and the progressive worsening of organ damage.

The physio-pathogenetic mechanisms of ischemic events in patients with SCD are numerous. Hypoxia conditions the formation of insoluble desoxy-Hb with consequent polymerization of HBS up to the formation of Hb (tactoids) gel. This generates: alteration and loss of elasticity of the erythrocyte membrane; formation of sickle and dence cells; alteration of the vascular endothelium. These events are the substratum of the pivotal mechanisms underlying the sickling crisis: hemolysis and vaso-occulsion.

Sickle cell disease is the most common hemoglobinopathy in Africa, the Middle East and the countries of Southeast Asia; the prevalence of SCD in Italy has significantly increased in recent years in relation to migratory flows from countries with high incidence of this disease.

In relation to Caritas data on immigration (1994 and 2000), an influx of about 10 new patients / year is expected. The ISTAT register, in 2010 in Lombardy the foreign population reached the incidence of 10.7% equal to 1064447, destined to increase over time; in particular Lombardy is the Italian region with the highest rate of immigrants (23.3%), followed by Lazio, Emilia Romagna and Veneto.

In 2006 the World Health Organization (WHO) called on governments to "formulate, implement, reinforce in a systematic way, fair and effective the national programs, global and integrated, for the prevention and treatment of sickle-cell disease in order to reduce mortality and morbidity" .

On 22/08/2008 the United Nations General Assembly established the World Sickle Disease Day.

In 2010 the WHO and the United Nations (www.afro.who.int) recognized the disease as a "global health problem".Based on the WHO recommendations and on the evidence of the increase in the number of patients seen in recent decades, also in relation to multiethnic migratory phenomena, the Italian Society of Thalassemia and Hemoglobinopathies (SITE), the Society Italian Transfusion Medicine and Immunohaematology (SIMTI) and the Italian Association of Hematology and Pediatric Oncology (AIEOP) have considered important to promote and propose a "Survey" that could allow to acquire information about the treatment, with particular regard to the transfusion therapy, offered to patients with sickle cell disease in the different Italian realities and at the same time perform a "mapping" of the Transfusion Structures that apply erythrocyte exchange programs. The resulting information can also constitute a valid and concrete help to the orientation of the patients themselves.

This is an observational study aimed to better understand the management criticalities of these patients (first of all difficulty in obtaining blood for different ethnic groups) and consisting in the acquisition of clinical and epidemiological data (age, ethnicity) on a national basis, referred to pediatric and adult patients. Patients included in the study will be able to refer to the total number of patients belonging to the Center, whether following a specific therapeutic program, or requiring no treatment and only in follow-up, in order to detect the overall number of patients.

The "Survey" is present online and accessible through the SITE website (www.SITE-italia.org) (initially, also via the sites of SIMTI and AIEOP), where it will be possible to find instructions for completing the collection form data, if the indications contained in the data sheet are not clear.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering of sickle cell disease, with diagnosis confirmed by standardized biochemical criteria or by matching mutations on globin genes by DNA analysis;
* all patients who consent to the study by signing the informed consent given by the U.O.C.

Exclusion Criteria:

* patients without a diagnosis confirmed according to standardized biochemical criteria or via mutation on globin genes by DNA analysis.
* all patients unable to understand the study protocol and to give informed consent and who have no legal representative.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All Survey participants will be recruited from the Centers distributed in Italy; inclusion in the study will be in compliance with the inclusion and exclusion criteria. The information and the manifestation of the Consent will be illustrated and, where necessary, discussed in the presence of a Cultural Linguistic Mediator.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Web-based recording of personal, therapy and complications data of patients with sickle cell anemia included in the National Transfusion Treatment Survey | Data will be recorded up to six months
  The Survey Data Sheet is divided into three parts:
  1. Personal data
  2. Therapy:
     * Chronic transfusion regimen
     * Acute transfusion regimen
     * Hydroxyurea
  3. Complications: -
     * Alloimmunization
     * Transfusion reactions
     * Martial structure and iron-chelating therapy

CONTACTS AND LOCATIONS:
Overall Officials: Giovanna Graziadei, MD, Principal Investigator — Fondazione IRCCS Policlinico di Milano con sede in Via Francesco Sforza 35, 20122 Milano
Locations (1):
- Gian Luca Forni, Genova, Ge, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ohene-Frempong K, Weiner SJ, Sleeper LA, Miller ST, Embury S, Moohr JW, Wethers DL, Pegelow CH, Gill FM. Cerebrovascular accidents in sickle cell disease: rates and risk factors. Blood. 1998 Jan 1;91(1):288-94. PMID 9414296
- [Background] Rees DC, Williams TN, Gladwin MT. Sickle-cell disease. Lancet. 2010 Dec 11;376(9757):2018-31. doi: 10.1016/S0140-6736(10)61029-X. Epub 2010 Dec 3. PMID 21131035
- [Background] Piel FB, Tatem AJ, Huang Z, Gupta S, Williams TN, Weatherall DJ. Global migration and the changing distribution of sickle haemoglobin: a quantitative study of temporal trends between 1960 and 2000. Lancet Glob Health. 2014 Feb;2(2):e80-9. doi: 10.1016/S2214-109X(13)70150-5. PMID 24748392
- [Background] Piel FB, Hay SI, Gupta S, Weatherall DJ, Williams TN. Global burden of sickle cell anaemia in children under five, 2010-2050: modelling based on demographics, excess mortality, and interventions. PLoS Med. 2013;10(7):e1001484. doi: 10.1371/journal.pmed.1001484. Epub 2013 Jul 16. PMID 23874164
- [Derived] Graziadei G, De Franceschi L, Sainati L, Venturelli D, Masera N, Bonomo P, Vassanelli A, Casale M, Lodi G, Voi V, Rigano P, Pinto VM, Quota A, Notarangelo LD, Russo G, Allo M, Rosso R, D'Ascola D, Facchini E, Macchi S, Arcioni F, Bonetti F, Rossi E, Sau A, Campisi S, Colarusso G, Giona F, Lisi R, Giordano P, Boscarol G, Filosa A, Marktel S, Maroni P, Murgia M, Origa R, Longo F, Bortolotti M, Colombatti R, Di Maggio R, Mariani R, Piperno A, Corti P, Fidone C, Palazzi G, Badalamenti L, Gianesin B, Piel FB, Forni GL. Transfusional Approach in Multi-Ethnic Sickle Cell Patients: Real-World Practice Data From a Multicenter Survey in Italy. Front Med (Lausanne). 2022 Mar 16;9:832154. doi: 10.3389/fmed.2022.832154. eCollection 2022. PMID 35372393